CLINICAL TRIAL: NCT02764840
Title: Muscular Resistance Test in the Elastic Tube: Reliability and Training of the Proposed Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: São Paulo State University (Other)
Responsible Party: Principal Investigator, Jaqueline Santos Silva, Master's Degree student, São Paulo State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SaoPSU
Record Dates: First submitted 2015-12-02; First posted 2016-05-06 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Muscle Strength Quantitative Trait Locus 1

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental group isokinetic dynamometer (GEDI) (Experimental): Isokinetic Biodex System Pro 4
  Interventions: Other: isokinetic dynamometer
- experimental group elastic tube (GETE) (Experimental): elastic tube brand LEMGRUBER 203
  Interventions: Other: elastic tube

INTERVENTIONS:
Other: isokinetic dynamometer — In the first stage a fatigue test will be applied. In the second stage, different participants will undergo a protocol for muscle strength gain. The first stage of the study will be crossover. The second will be split, one arm carry out the procedures in the elastic tube and the other in isokinetic dynamometer.
  Arms: experimental group isokinetic dynamometer (GEDI)
Other: elastic tube — In the first stage a fatigue test will be applied. In the second stage, different participants will undergo a protocol for muscle strength gain.
  Arms: experimental group elastic tube (GETE)

SUMMARY:
Resistance exercises from elastic tube has been used as part of the rehabilitation and maintenance of muscle tone levels in different scenarios, from disease conditions to the sports universe. There is the convenience and low cost of the instrument, which can provide impact on clinical and economic framework in case of spillage of use strategies. In a recent search, the investigators were not observed data on the reliability and reproducibility of a specific test for this tool and in this sense, it seems pertinent to undertake research on the topic. Objectives: To determine the reliability and reproducibility by comparison with a isokinetic muscle strength test located â fatigue held in elastic tube and compare the results of a training protocol for muscle strength gain in both methods, elastic tube and dynamometer. Methods: Participants will perform the muscular endurance test localized fatigue, on two occasions, with an interval of seven days between them. Everyone will accomplish so much in the elastic tube, as in the isokinetic dynamometer. It will be held evaluator analysis intra and inter evaluator. After first stage of the study to determine the reliability test, the participants will undergo three weeks of training to gain muscular endurance, distributed in two groups G1 (training in the elastic tube) and G2 (training in isokinetic dynamometer) previously randomized. It will use the intra-class correlation coefficient with 95% confidence interval to check the repeatability and the Kappa coefficient with 95% confidence interval for reproducibility. To compare the responses of training, the distribution will be made as to the normality of the data by the Kolmogorov-Smirnov test. In the case of normal distribution, the Student's t-test for unpaired data and Mann-Whitney will be adopted if there is no normal distribution.

DETAILED DESCRIPTION:
The objectives of this study are: to assess the reliability of a method fatigue resistance assessment with elastic tube in two areas, inter and intra-examiner; check test reproducibility at different times with the same participant and compare this method with the gold standard of evaluation, the isokinetic dynamometer and compare the strength gains and endurance after the application of specific training in the elastic tube and an isokinetic dynamometer. It is a study of reproducibility, followed by application of a training protocol featuring a clinical trial.

Data collection will be held at the Center for Studies and Assistance in Physical Therapy and Rehabilitation (CEAFIR) FCT / UNESP, respecting the hours of 17:00 to 22:00. The study will be conducted in two stages: Reliability and reproducibility, and Training.

In the first stage of the study, the procedures will be conducted in six sessions. In the first, participants will be submitted to anthropometric measurements, questionnaires on physical activity level (IPAQ and Baecke) Contraction Maximum Voluntary (CVM) in isokinetic dynamometer test familiarization in the first analysis tool (elastic tube or isokinetic dynamometer) previously randomized. Randomization will be made by lot in Excel. It will be given interval of two days between the familiar and the first test.

In the second session, participants will perform the same test twice, with standardized interval of five minutes. In each test there will be a different supervisory therapist order to check whether or not the correlation between therapists.

In the third session, seven days after the initial tests, retests will be carried out by the same therapists who oversaw the previous session, aimed at finding or non-compliance of the information recorded in each of the therapists. In fitness tests, a seven-day period of separation is commonly used. For both the test will be played on two occasions separated by seven days.

In order to control possible biases, the order of application of the assessors in the test and retest will be crossed, and the first evaluating the test, shall be according reviewer on retest and vice versa. Furthermore, in all test sessions, it is inserted after the application of the first evaluator, a five minute rest and after, application of a Likert scale recovery Perception before the second evaluator start the test. If the participant reports of less than seven, it is understood that is not yet recovered and in these cases the scale is reapplied at intervals of one minute until the reported value exceeds seven. The choice of value is based on a priori knowledge acquired by pilot and respects the biological individuality of the participant. Although this age group and the sample health conditions non-recovery situations are exceptions, it is understood that the disposal of information is not adequate as far as the individual profile of each participant recovery. As the central object in this case is the test, it is the option for ensuring the inclusion of eligible study and use of the information with greater control of background levels of the participants. Such information is logged for further discussion. Tests conducted in both tools will be preceded by a warming of ten repetitions of knee flexion-extension of the dominant limb without charge.

Finalized the procedures in the first tool, the participants will undergo cross, starting in the fourth, fifth and sixth session procedures identical to the first three sessions, differing only the tool. This stage of the study will be cross over In the second stage of the study, the sample is again randomized and allocated to two groups (G1 and G2). The periodization of the groups will be identical, differing from the instrument and its features, which will be outlined in procedures.

ELIGIBILITY:
Inclusion Criteria:

* healthy young and physically active

Exclusion Criteria:

* be alcoholic, drug use, smoking or anti-inflammatory drugs chronically, present anemia, inflammation, diabetes, cardiovascular disease, liver problems and episode of muscle-tendon or osteo-articular lesions in the lower limbs and / or spine in the last six months

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 230 (Actual)
Dates: Start 2015-02; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Reliability of the proposed test | up to four weeks
  In the first stage of the study analyzes will be performed to evaluate test reliability. Measurements will be performed on the isokinetic dynamometer, and measures shall be given in Nm

SECONDARY OUTCOMES:
measure the gain endurance and strength | up to four weeks
  In the second stage of the study participants will undergo a training protocol to gain muscle strength. The primary outcome measure is the resistance and secondary force.Measurements will be performed on the isokinetic dynamometer, and measures shall be given in Nm

CONTACTS AND LOCATIONS:
Overall Officials: Jaqueline Silva, student, Principal Investigator — São Paulo State University
Locations (1):
- Paulista State University, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes